CLINICAL TRIAL: NCT00913653
Title: An Open Label, Non-randomised Study to Explore Safety/Tolerability, Pharmacokinetics and Pharmacodynamics of LCZ696 in Patients With Stable Heart Failure
Brief Title: Safety/Tolerability, Pharmacokinetics/Pharmacodynamics (PK/PD) of LCZ696 in Patients With Stable Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696A2117
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-11

CONDITIONS: Heart Failure
Keywords: Heart failure; LCZ696
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stable heart failure patients (Experimental)
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696

SUMMARY:
This study assess the safety/tolerability, PK/PD of LCZ696 in patients with stable heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented heart failure (NYHA class II-IV)

Exclusion Criteria:

* Use of both ACEi and ARB, ACEi and DRI, ARB and DRI treatment, or all three medications at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety (including blood pressure, renal function and serum electrolytes) and tolerability of LCZ696 | 14 days

SECONDARY OUTCOMES:
Pharmacokinetics of LCZ696 and its metabolites | 14 days
Pharmacodynamics of LCZ696 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- GOUVPO Russian Peoples´ Friendship University, Center of Applied, Moscow, Russia

REFERENCES:
- [Result] Kobalava Z, Kotovskaya Y, Averkov O, Pavlikova E, Moiseev V, Albrecht D, Chandra P, Ayalasomayajula S, Prescott MF, Pal P, Langenickel TH, Jordaan P, Rajman I. Pharmacodynamic and Pharmacokinetic Profiles of Sacubitril/Valsartan (LCZ696) in Patients with Heart Failure and Reduced Ejection Fraction. Cardiovasc Ther. 2016 Aug;34(4):191-8. doi: 10.1111/1755-5922.12183. PMID 26990595
- See also: Results for CLCZ696A2117 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3202